CLINICAL TRIAL: NCT03237299
Title: Loco-regional Complications of Pharyngitis in Children: a National Case-Control Study
Acronym: CAPE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI14034J
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Pharyngitis
Keywords: Pharyngitis; case-control study; loco-regional complications of pharyngitis
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases: children with loco-regional complications of pharyngitis
  Interventions: Other: Collection of data
- Controls: Controls: children with pharyngitis but without infectious complications
  Interventions: Other: No collection of data

INTERVENTIONS:
Other: Collection of data — Collection of data on clinical, bacteriological and computed tomography data concerning the case, which will be needed by the adjudication committee and for defining the index date.
  Groups: Cases
Other: No collection of data — The interviewer will note sociodemographic characteristics (age, weight, sex), symptoms and their evolution, and all drug intakes of the patient during the month before the index date.
  Groups: Controls

SUMMARY:
To study the association between several exposures of interest and the occurrence of infectious loco-regional complications of pharyngitis in children.

DETAILED DESCRIPTION:
Investigators will include in the study (after agreement of child and parents):

* Cases: children < 18 years old hospitalized for peripharyngeal suppurations, diffuse cervical cellulitis or cervical adenophlegmon in participating Ear, Nose & Throat (ENT) and pediatric departments.
* Controls: children < 18 years old with pharyngitis but without infectious complications recruited by general practitioners (GPs) or by primary care pediatricians in private setting, matched to cases by age, date of infectious complication (index date), delay between the pharyngitis and the index date and, if possible, the referring physician.

Primary endpoint: Difference in the frequency of exposure to various factors among cases and controls during an exposure window going from the date of diagnosis of pharyngitis to day -0.5 of the index date of the complication.

Several exposure of interest will be compared between cases and controls. One specific main exposure of interest during a predefined window of exposure has been defined but will not be revealed to investigators to avoid selection bias. Several secondary exposure of interest were a priori defined but will not be revealed to investigators to avoid selection bias.

ELIGIBILITY:
Inclusion Criteria:

Cases: children < 18 years old hospitalized for peripharyngeal suppurations, diffuse cervical cellulitis or cervical adenophlegmon in participating Ear, Nose & Throat (ENT) and pediatric departments.

Controls: children < 18 years old with pharyngitis but without infectious complications recruited by general practitioners (GPs) or by primary care pediatricians in private setting, matched to cases by age, date of infectious complication (index date), delay between the pharyngitis and the index date and, if possible, the referring physician.

Exclusion Criteria:

Children (cases or controls) with chronic renal failure, hemophilia, chronic thrombocytopenia or immunosuppression (constitutional or iatrogenic) at the time of pharyngitis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cases: participating Ear, Nose & Throat (ENT) and pediatric departments Controls: recruited ''in office settings'' by general practitioners (GPs) or by primary care paediatricians
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Frequency of exposure of interest | from the date of diagnosis of pharyngitis up to 6 weeks

SECONDARY OUTCOMES:
Magnitude of the exposure of interest | from the date of diagnosis of pharyngitis up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin CHALUMEAU, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants Malades - AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: No